CLINICAL TRIAL: NCT04843449
Title: A Phase I, Open Label, Drug-drug Interaction Study to Evaluate the Effects of Itraconazole and Rifampin on the Pharmacokinetics of ASC40 in Healthy Subjects
Brief Title: Study to Evaluate the Effects of Itraconazole and Rifampin on the Pharmacokinetics of ASC40 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASC40-102
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Healthy Volunteers; DDI (Drug-Drug Interaction); Itraconazole; Rifampicin; ASC40
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitor group (Experimental): 1. ASC40 50mg, once daily on the 1st and 11th days before meal;
  2. Itraconazole 200mg, once daily from the 6th day to the 15th day.
  Interventions: Drug: ASC40; Drug: Itraconazole
- Inducer group (Experimental): 1. ASC40 50mg, once daily on the 1st and 19th days before meal;
  2. Rifampicin 600mg, once daily from the 6th day to the 19th day.
  Interventions: Drug: ASC40; Drug: rifampicin

INTERVENTIONS:
Drug: ASC40 — Oral tablets
Drug: Itraconazole — Oral capsules
  Arms: Inhibitor group
Drug: rifampicin — Oral capsules
  Arms: Inducer group

SUMMARY:
The primary objective of this study is to evaluate the effects of itraconazole (a strong inhibitor of cytochrome P450 3A (CYP3A)) and rifampicin (a strong inducer of CYP3A) on the pharmacokinetics of ASC40 in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

-19kg/m2 ≤ BMI <40kg/m2.

Key Exclusion Criteria:

* History of, or current digestive system, nervous system disease, etc..
* Taking drugs or foods that inhibit or induce the liver's metabolism.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
AUC of ASC40 | Up to 24 days
  Evaluate the Area under the Plasma Concentration Versus Time Curve after single oral dose of ASC40 administered to healthy volunteers in the presence or absence of CYP3A inhibitor or inducer.
Cmax of ASC40 | Up to 24 days
  Evaluate the Peak Plasma Concentration after single oral dose of ASC40 administered to healthy volunteers in the presence or absence of CYP3A inhibitor or inducer.

SECONDARY OUTCOMES:
t1/2 of ASC40 | Up to 24 days
  Evaluate the Terminal-Phase Half-Life after single oral dose of ASC40 administered to healthy volunteers in the presence or absence of CYP3A inhibitor or inducer.
CL/F of ASC40 | Up to 24 days
  Evaluate the Apparent Systemic Clearance after single oral dose of ASC40 administered to healthy volunteers in the presence or absence of CYP3A inhibitor or inducer.
Vd/F of ASC40 | Up to 24 days
  Evaluate the Apparent Volume of Distribution after single oral dose of ASC40 administered to healthy volunteers in the presence or absence of CYP3A inhibitor or inducer.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 24 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan provincial people's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided